CLINICAL TRIAL: NCT03509376
Title: Operative Correction of Abdominal Rectus Diastasis (ARD): the Effect on Low Back Pain and Movement Control. A Randomized, Prospective Trial Comparing Novel, Mini-invasive Mesh Repair to Plication
Brief Title: Operative Correction of Rectus Muscle Diastasis (ARD): the Effect on Low Back Pain and Movement Control
Acronym: RmB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: Oulu University Hospital (Other)
Responsible Party: Principal Investigator, Jaana Vironen, Chief surgeon, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUS/26/2018
Record Dates: First submitted 2018-04-11; First posted 2018-04-26 (Actual); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Diastasis Recti

STUDY DESIGN:
Intervention Model Description: Patients are randomised to a suture repair or suture with mesh repair
Who Masked: Outcomes Assessor
Masking Description: The physiotherapist doing the clinical examinations at different phases of the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Suture repair (Experimental): Diastasis recti is repaired using nylon suture for the plication
  Interventions: Procedure: Suture repair
- Rolled mesh repair (Experimental): Diastasis recti is repaired with self gripping mesh to reinforce the suture line
  Interventions: Procedure: Rolled mesh repair

INTERVENTIONS:
Procedure: Suture repair — The diastasis is repaired with continous nylon suture
  Arms: Suture repair
Procedure: Rolled mesh repair — Continuous nylon suture is done over a narrow strip of self gripping Rolled mesh to repair the diastasis
  Arms: Rolled mesh repair

SUMMARY:
This study is a randomized controlled trial comparing two ADR repair methods: nylon suturing and nylon suture with mesh enforcement. The ADR correction is performed simultaneously with abdominoplasty/ modified skin reduction abdominoplasty.

DETAILED DESCRIPTION:
Abdominal diastasis recti (ADR) persists after pregnancies in one third of women. Traditionally plain ADR has been managed conservatively. There is some evidence that ADR reduces abdominal integrity and functional strength, contributing to pelvic instability and back pain. However, patients are referred to a surgeon mainly because of some other primary concern and ADR is an additional condition: in the case of excess skin-subcutis, the person is referred to a plastic and reconstructive surgeon for abdominoplasty and in the case of midline hernia, to a general surgeon.

In combination with abdominoplasty the plication of the superficial aponeurosis of recti muscles is the most commonly used reconstructive technique. There is a wide variety of different plication procedures available. Convincing data of the long-term results of ADR repair are lacking especially when ADR is severe. Some studies have reported large recurrence rates. Polypropylene mesh repair is an evidence-based technique to ensure a strong and reliable abdominal wall repair in ventral hernias or in high risk laparotomy wounds. Large retromuscular or intraperitoneal meshes have been used also in ARD repair.

This study reports a novel surgical technique aimed at reliable and mini-invasive open repair of ADR with or without midline hernia combined by abdominoplasty for symptomatic ADR patients. In RmB (roll mesh in between) method the investigators bury a narrow piece of self-gripping mesh inside the plicated linea alba to give tensile strength to plication. Patients are randomized to a suture plication group or RmB group.

Outcome evaluation is performed by clinical examination with video recorded movement control tests and with structured questionnaires for Quality of Life (RAND36) and for low back pain (LBP) (Oswestry 2.0). Evaluation is done three times: when recruiting the patient, after a conservative 3-6 months therapy with written instructions and one year after the intervention. Complications and recurrences are recorded as well.

Outcomes The effect of ADR repair on LBP and movement control problems Patient satisfaction and complications of ADR repair after the two techniques

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic diastasis recti (> 3 cm) after pregnancies, with or without a midline hernia

Exclusion Criteria:

* BMI > 28,
* smoking
* less than a year since the previous pregnancy or still breast feeding
* planning further pregnancies

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Low back pain | At one year
  Improvement in Oswestry 2.0 score

SECONDARY OUTCOMES:
Recurrence | at 1 year
  Number of symptomatic, recurrent diastasis > 3 cm
Quality of life | at one year
  RAND 36 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Tiina Jahkola, Principal Investigator — Helsinki University Central Hospital; Tero Rautio, Principal Investigator — Oulu University Hospital; Katariina Kilpivaara, Principal Investigator — Oulu University Hospital
Locations (2):
- Finland (2):
  - HUCH Jorvi Hospital, department of Surgery, Espoo
  - Oulu University Hospital, Oulu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tuominen R, Saxen J, Jahkola T, Mikkonen J, Arokoski J, Luomajoki H, Vironen J. Rectus diastasis repair with and without mesh at 1 year: randomized clinical trial. Br J Surg. 2025 Nov 6;112(11):znaf231. doi: 10.1093/bjs/znaf231. PMID 41289051